CLINICAL TRIAL: NCT04626427
Title: The WavelinQ™ Arterio-Venous Endovascular Fistula: A Global, Multi-Center, Prospective, Post-Market, Confirmatory, Interventional, Investigation
Brief Title: The WavelinQ™ Arterio-Venous Endovascular Fistula: A Global, Post-Market Investigation
Acronym: WAVE-Global
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to shifting post-pandemic clinical landscape, concurrent study (NCT04634916) to provide results on analogous endpoints in advance of current projections
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDPI-19-005
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-03

CONDITIONS: End Stage Kidney Disease; Chronic Kidney Diseases; Kidney Failure; Kidney Insufficiency; Kidney Disease, Chronic; AV Fistula; Fistulas Arteriovenous
Keywords: Kidney Replacement Therapy; Hemodialysis; Vascular Access; Arteriovenous Access; Arteriovenous Fistula; Endovascular Arteriovenous Fistula
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Renal Insufficiency; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- WavelinQ™ EndoAVF System (Experimental): The WavelinQ™ EndoAVF System is indicated for the cutting and coagulation of blood vessel tissue in the peripheral vasculature for the creation of an AVF used for HD. The device is intended to be used in patients suffering from chronic kidney disease requiring HD by physicians trained and experienced in endovascular techniques. The WavelinQ™ EndoAVF System will be used for these intended purposes as part of this clinical investigation according to its instructions for use (IFU).
  Interventions: Device: WavelinQ™ EndoAVF System

INTERVENTIONS:
Device: WavelinQ™ EndoAVF System — AVF endovascular creations using the WavelinQ™ EndoAVF System

SUMMARY:
This is a global, multi-center, prospective, post-market, confirmatory, interventional, non-randomized, single-arm clinical investigation evaluating arteriovenous fistula (AVF) creation by means of the WavelinQ™ EndoAVF System in patients who require a vascular access for hemodialysis (HD).

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to provide clinical evidence to further demonstrate reasonable assurance of safety and effectiveness of the WavelinQ™ EndoAVF System when used for endovascular arteriovenous fistula (endoAVF) creations. Treated participants will be followed for 24-months post index procedure.

ELIGIBILITY:
Inclusion Criteria:

The participant must:

1. Be able to comprehend, voluntarily sign and date the informed consent form (ICF) prior to collection of clinical investigation data or performance of clinical investigation procedures (or where allowable the participant's legally authorized representative (LAR) on behalf of the participant).
2. Be able to and willing to comply with the CIP requirements, including clinical follow-up.
3. Be male or non-pregnant female ≥ 18 years of age with an expected lifespan sufficient (≥ 24 months) to allow for completion of all clinical investigation procedures.
4. Have established, non-reversible kidney failure, who are currently on HD at screening or are in need of a vascular access for HD as determined by the referring clinician.
5. Target treatment vein diameter(s) for AVF creation ≥ 2.0 mm as measured via DUS or angiography.
6. A target treatment artery diameter ≥ 2.0 mm as measured via DUS or angiography.
7. Adequate collateral circulation to the hand, in the opinion of the Principal Investigator (PI) (or authorized designee).
8. At least one superficial outflow vein diameter ≥ 2.5 mm as measured via DUS or angiography that is in communication with the target creation site via a proximal forearm perforating vein.

Exclusion Criteria:

The participant must not have:

1. Active or nontreated hypercoagulable state.
2. Known bleeding diathesis.
3. Insufficient cardiac output to support the maturation and use of an AVF in the opinion of the PI (or authorized designee).
4. Known history of or current active intravenous drug abuse.
5. A "planned" major surgical procedure within 6 months following index procedure or major surgery, in the opinion of the PI (or authorized designee), within 30 days prior to index procedure.
6. Known allergy or hypersensitivity to contrast media which cannot be adequately treated with pre-medication.
7. Known adverse effects to sedation and / or anesthesia which cannot be adequately treated with pre-medication.
8. Evidence of active infection on the day of the index procedure (temperature of ≥ 38.0° Celsius and / or White Blood Cell (WBC) Count of ≥ 12,000 cells / μL, if collected).
9. Another medical condition, which, in the opinion of the PI (or authorized designee), may cause him / her to be non-compliant with the CIP, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of clinical investigation procedures and follow-up.
10. Current participation in an investigational drug or device clinical investigation that has not completed the clinical investigation treatment or that clinically interferes with the clinical investigation endpoints. Note: Investigations requiring extended follow-up visits for products that were investigational, but have since become commercially available, are not considered investigational.
11. Central venous stenosis or central vein narrowing ≥ 50% based on imaging, or any degree of central venous stenosis with accompanying signs or symptoms, on the same side as the planned AVF creation.
12. The absence of a proximal forearm perforating vein feeding the target cannulation vein(s) from the target creation site via DUS or angiography.
13. Occlusion or stenosis ≥ 50%, or any degree of stenosis with accompanying signs or symptoms of target cannulation vein(s) such as cephalic, median cubital, basilic, etc. assessed via DUS or angiography and as clinically determined by PI (or authorized designee).
14. Significantly compromised venous or arterial architecture (e.g. severe vessel calcification) or flow in the treatment arm as determined by the PI (or authorized designee) and DUS or angiography.
15. Presence of significant calcification at the target endoAVF location that could potentially impact the effectiveness of endoAVF creation as determined by the PI (or authorized designee).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charmaine Lok, MD, MSc, Principal Investigator — University Health Network, Toronto; Nicholas Inston, PhD, Principal Investigator — The Queen Elizabeth Hospital; Panagiotis Kitrou, MD, MSc, PhD, Principal Investigator — University Hospital of Patras
Locations (3):
- Imelda Hospital Bonheiden, Bonheiden, Belgium
- University Hospital of Patras "Panagia I Voitheia", Rio, Greece
- Kantonsspital Winterthur, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 participants signed informed consent prior to investigation early termination.
Pre-assignment Details: 21 participants had signed informed consent. 14 were treated with the device. Six (6) were screen failures: Four (4) did not meet anatomical eligibility and two (2) did not meet clinical eligibility criteria. One (1) participant did not have the device inserted. This participant had signed consent prior to investigation termination but the procedure was completed after the investigation had terminated as part of standard of care.
Groups:
- WavelinQ™ EndoAVF System: The WavelinQ™ EndoAVF System is indicated for the cutting and coagulation of blood vessel tissue in the peripheral vasculature for the creation of an arteriovenous fistula (AVF) used for hemodialysis (HD). The device is intended to be used in patients suffering from chronic kidney disease requiring HD by physicians trained and experienced in endovascular techniques. The WavelinQ™ EndoAVF System was used for these intended purposes as part of this clinical investigation according to its instructions for use (IFU).
  WavelinQ™ EndoAVF System: AVF endovascular creations using the WavelinQ™ EndoAVF System
Period: Overall Study
Arm/Group | WavelinQ™ EndoAVF System
Started | 14
30-Day Follow-Up | 13
6-Week Follow-Up | 12
3-Month Follow-Up | 12
6-Month Follow-Up | 11
12-Month Follow-Up | 2
Completed | 0
Not Completed | 14
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Investigation Early Termination by Sponsor | 11
Not completed — Participant Permanently Moved Abroad | 1

BASELINE CHARACTERISTICS:
Arm/Group | WavelinQ™ EndoAVF System
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (16.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Greece | 5
  Belgium | 5
  Switzerland | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.91 (4.536)

OUTCOME MEASURES:

1. Primary Outcome: Safety: Device and Procedure Related Serious Adverse Events (SAEs) - Presented as the Number of Participants With Freedom From Clinical Events Committee (CEC) Adjudicated Device and/or Procedure-Related SAEs.
Description: Clinical Investigation Plan (CIP) Endpoint Definition: The proportion of participants with freedom from CEC adjudicated device- or procedure-related SAEs.
  The CEC established criteria to determine the relatability of an adverse event (AE) to the device and/or the index procedure. Based on these criteria, AEs were adjudicated to be "definitely related", "possibly related", or "not related". Events adjudicated to be "definitely" or "possibly" related were considered to be related events.
  NOTE: Due to early termination of the investigation, this endpoint is presented as the number of participants with freedom from CEC adjudicated device- or procedure-related SAEs.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- WavelinQ™ EndoAVF System: The WavelinQ™ EndoAVF System is indicated for the cutting and coagulation of blood vessel tissue in the peripheral vasculature for the creation of an AVF used for HD. The device is intended to be used in patients suffering from chronic kidney disease requiring HD by physicians trained and experienced in endovascular techniques. The WavelinQ™ EndoAVF System was used for these intended purposes as part of this clinical investigation according to its IFU.
  WavelinQ™ EndoAVF System: AVF endovascular creations using the WavelinQ™ EndoAVF System
Arm/Group | WavelinQ™ EndoAVF System
Number analyzed (Participants) | 13
Participants
  Overall Number of Participants with Freedom from CEC Adjudicated Device &/ Procedure Related SAEs | 12
  Possible Procedure-Related SAE (Azotaemia - 7 days Post-Index Procedure with 4 Day Hospitalization) | 1

2. Primary Outcome: Effectiveness: Number of Interventions Per Patient Years to Facilitate and / or Maintain AVF Use
Description: CIP Endpoint Definition: The number of interventions per patient years to facilitate and / or maintain AVF use (facilitation interventions and / or maintenance interventions). The assessment of interventions to facilitate and/or maintain AVF use started post creation (after the completion of the index procedure).
  NOTE: For the calculation of the endpoint, the number of Interventions per Patient Years to Facilitate and / or Maintain AVF Use was to be estimated by using the Poisson regression model. Given the early termination of the investigation the mean and standard deviation of the Number of Interventions and Patient Years used for the derivation are provided in the Analysis Population Description.
Time Frame: 6 months
Population: To provide details on the calculation on the rate given the early termination of the investigation - the mean (standard deviation) number of interventions used was 0.5 (0.76) and the mean (standard deviation) number of patient years used was 0.5 (0.20). This provided the rate presented in the Outcome Measure Data Table.
Measure: Number; unit: Number of Interventions / Patient Years
Arm/Group | WavelinQ™ EndoAVF System
Number analyzed (Participants) | 14
Number of Interventions / Patient Years | 1.00

3. Secondary Outcome: Device and Procedure Related SAEs - Presented as the Number of Participants With Freedom From CEC Adjudicated Device and/or Procedure-Related SAEs.
Description: CIP Endpoint Definition: The proportion of participants with freedom from CEC adjudicated device- or procedure-related SAEs.
  The CEC established criteria to determine the relatability of an adverse event (AE) to the device and/or the index procedure. Based on these criteria, AEs were adjudicated to be "definitely related", "possibly related", or "not related". Events adjudicated to be "definitely" or "possibly" related were considered to be related events.
  NOTE: Due to early termination of the investigation, this endpoint is presented as the number of participants with freedom from CEC adjudicated device- or procedure-related SAEs. This included the assessment of the 12 participants that reached 6-months prior to investigation early termination. No further related SAEs were identified in this time period from the one part of the primary safety endpoint.
Time Frame: 6 months (24 months was also to be reported per the CIP but due to investigation early termination only data through 6 months was able to be evaluated).
Measure: Count of Participants; unit: Participants
Arm/Group | WavelinQ™ EndoAVF System
Number analyzed (Participants) | 12
Participants
  Overall Number of Participants with Freedom from CEC Adjudicated Device &/ Procedure Related SAEs | 11
  Possible Procedure-Related SAE (Azotaemia - 7 days Post-Index Procedure with 4 Day Hospitalization) | 1

4. Secondary Outcome: Physiological Maturation - Presented as the Number of Participants With AVFs That Meet the CIP Definition of Physiological Maturation as Measured by Duplex Ultrasound (DUS).
Description: CIP Endpoint Definition: The proportion of participants with AVFs that meet the CIP definition of physiological maturation as measured by DUS. Core Lab data was the primary source for endpoint derivation. In the event where core lab data was unavailable, site reported data was used.
  Physiological maturation was defined as an AVF having at least 500 mL/min of flow in the brachial artery and an outflow vein diameter of ≥4 mm as measured by DUS. Participants with AVFs that met the definition of functional maturation were automatically considered to have met the endpoint of physiological maturation.
  NOTE: Due to the early termination of the investigation this endpoint is presented as the number of participants with AVFs that meet the definition of physiological maturation as measured by DUS.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | WavelinQ™ EndoAVF System
Number analyzed (Participants) | 13
Participants
  Overall Number of Participants with Physiological Maturation | 12
  Missing DUS / HD Data - Unable to Confirm Physiological Maturation (CIP Deviation) | 1

5. Secondary Outcome: Cannulation Success - Presented as the Percentage of Participants With Cannulation Success.
Description: CIP Endpoint Definition: The interval of time between HD arteriovenous (AV) access creation to first successful use for HD and proportion of participants with successful first use for HD as defined in the CIP. Cannulation Success is defined as the first successful use for HD using 2-needle cannulation.
  NOTE: Given the early termination of the investigation, this endpoint is presented as the percentage of participants with successful first use for HD. The Kaplan-Meier (KM) method was used to estimate the proportion of participants with success at 6 months.
Time Frame: 6 months
Population: NOTE: The overall assessment of the fourteen (14) participants includes three (3) incident (pre-HD) participants that never required HD during the investigation. The % of the eleven (11) subjects that were eligible for HD during the course of the investigation that achieved cannulation success prior to investigation early termination is also provided in the outcome table.
Measure: Number; unit: % of Participants with Success
Arm/Group | WavelinQ™ EndoAVF System
Number analyzed (Participants) | 14
% of Participants with Success
  Percentage of All Participants with Success - KM (%) | 46.2
  Percentage of HD Eligible Participants with Cannulation Success (%): number analyzed (Participants) | 11
  Percentage of HD Eligible Participants with Cannulation Success (%) | 72.7

6. Secondary Outcome: Cannulation Success - Presented as the Number of Days to Cannulation Success.
Description: CIP Endpoint Definition: The interval of time between HD arteriovenous (AV) access creation to first successful use for HD and proportion of participants with successful first use for HD as defined in the CIP. Cannulation Success is defined as the first successful use for HD using 2-needle cannulation. The median time to success was to be estimated using the Kaplan Meier curve and defined as the time at which 50% of participants reached success by the end of the 6-month window. By the end of the 6-month window, the estimated success rate was 46.2% (see Secondary Outcome above "Cannulation Success - Percentage of Participants With Cannulation Success") as such, there weren't sufficient data points with successes to get this estimate. Instead the minimum and maximum number of days to cannulation success for all participants through investigation early termination is provided.
Time Frame: Through Investigation Early Termination
Population: NOTE: The overall assessment of the fourteen (14) participants includes three (3) incident (pre-HD) participants that never required HD during the investigation.
Measure: Median (Full Range); unit: Time to Success (Days)
Arm/Group | WavelinQ™ EndoAVF System
Number analyzed (Participants) | 14
Time to Success (Days) | NA [32 to 210] — Given the definition of the median time to success (see "Outcome Measure Description") and the limited sample size due to early termination this estimate could not be determined.

7. Secondary Outcome: Cumulative Functional Patency - Presented as the Number of Participants With Cumulative Functional Patency
Description: CIP Endpoint Definition: The time from first successful HD AV access use for HD using 2-needle cannulation to access abandonment, when the access reaches an access censoring event as specified a priori in the CIP, or analysis timepoint / clinical investigation end.
  NOTE: Given the early termination of the investigation the endpoint is presented as the number of participants that had met the definition of cumulative functional patency - those that (1) had initiated HD successfully through their AVF with 2-needle cannulation and (2) whose AVF was not abandoned.
Time Frame: 6 months (12 months per CIP but due to investigation early termination data is reported through 6 months instead due to the limited resultant data available at 12 months)
Population: For the five (5) participants that had sufficient follow-up time prior to investigation termination, the cumulative functional patency through 6-months was evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | WavelinQ™ EndoAVF System
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Per the CIP, Adverse Events (AEs) were to be collected for intent-to-treat (ITT) participants immediately following the start of the index procedure (defined to start at the time of the initial skin puncture to gain vessel access) for the entire follow-up period of 24 months. Given the early termination of the investigation, the time frame varied individually for each participant - the mean number of years of follow up (standard deviation) was 0.498 (0.2).
Description: ISO14155:2020 definitions were used for adverse events (AEs) and serious adverse events (SAEs). Note: Planned hospital visits and / or hospital stays, or procedures required by the CIP (including subsequent interventions assessed in the clinical investigation endpoints), without serious deterioration in health were not to be considered SAEs.
Arm/Group | WavelinQ™ EndoAVF System
All-Cause Mortality (participants affected / at risk) | 1/14
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WavelinQ™ EndoAVF System (N=14)
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 1 (3) — Mid Cubital Post Surgical Vein Stenosis - Day 152, Day 203 and Day 256 - Not Related to Device or Procedure; Definitely Related to AV Access Circuit.
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 1 (1) — Ulnar Vein Stenosis - Day 245 - Not Related to Device or Procedure; Definitely Related to AV Access Circuit.
Arteriovenous Fistula Site Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) — Anastomosis Ulnar Site: Pseudoaneurysm - Day 373 - Possibly Related to Device and Procedure; Definitely Related to AV Access Circuit.
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 1 (1) — Anastomosis Ulnar Site: Thrombosis - Day 373 - Possibly Related to Device and Procedure; Definitely Related to AV Access Circuit
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 1 (1) — Stenosis Basilic Vein - Day 185 - Not Related to Device or Procedure; Definitely Related to AV Access Circuit
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Carcinoma - Day 216 - Not Related to Device, Procedure or AV Access Circuit.
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 1 (1) — Stenosis In Left Radial Vein - Day 218 - Not Related to Device or Procedure; Definitely Related to the AV Access Circuit.
Azotaemia (Renal and urinary disorders) | 1 (1) — Worsening Renal Function - Aggravated Pre-Existing Uremia - Day 8 - Not Related to Device; Possibly Related to Procedure; Not Related to AV Access Circuit.
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 1 (1) — Stenosis Between Vena Perforans and Vena Cephalica, Right Arm - Day 120 - Not Related to Device or Procedure; Definitely Related to AV Access Circuit
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 1 (1) — Stenosis Left Arm Perforator Vein - Day 136 - Not Related to Device or Procedure; Definitely Related to AV Access Circuit
Staphylococcal Sepsis (Infections and infestations) | 1 (1) — Infection With Staphylococcus Aureus - Sepsis - Day 145 - Not Related to Device, Procedure, or AV Access Circuit
Brachiocephalic Vein Stenosis (Vascular disorders) | 1 (1) — Stenosis Vena Brachiocephalica Left - Day 163 - Not Related to Device or Procedure; Definitely Related to AV Access Circuit
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WavelinQ™ EndoAVF System (N=14)
Puncture Site Haematoma (General disorders) | 1 (1) — Mild Hematoma - Day 1 - Not Related to Device; Definitely Related to Procedure and AV Access Circuit
Covid-19 (Infections and infestations) | 1 (1) — Covid-19 - Day 298 - Not Related to Device, Procedure, or AV Access Circuit
Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) — Fracture Dig. V, Left Hand - Day 164 - Not Related to Device, Procedure, or AV Access Circuit
Catheter Site Haemorrhage (General disorders) | 1 (1) — Seeping Hemorrhage Palindroma Catheter Right - Day 163 - Not Related to Device, Procedure, or AV Access Circuit

LIMITATIONS AND CAVEATS:
Early termination leading to small number of participants analyzed. Given the limited sample size of the investigation population, the testing of the hypotheses described in the CIP was not completed for the primary endpoints and instead data are presented in a descriptive fashion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT04626427/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT04626427/SAP_001.pdf